CLINICAL TRIAL: NCT07359625
Title: KETO-SENSE - Effects of Ketone Bodies on Insulin Sensitivity
Brief Title: Effects of Ketone Bodies on Insulin Sensitivity
Acronym: KETO-SENSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: KETO-SENSE
Record Dates: First submitted 2025-11-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Insulin Resistance; Obesity & Overweight; Energy Metabolism; Ketone Body Metabolism
Keywords: insulin resistance; Overweight; Growth hormone; Ketone bodies; Lipolysis; Energy metabolism
MeSH Terms: conditions — Insulin Resistance; Obesity; Overweight | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GH infusion + oral ketone supplement (Experimental): Participants receive a continuous intravenous infusion of growth hormone (30 ng·kg-¹·min-¹) combined with oral ketone supplementation.
  Interventions: Drug: Growth Hormone, Human; Dietary Supplement: Oral ketone supplement (KetoAid®, KE4)
- GH infusion + oral placebo (Experimental): Participants receive a continuous intravenous infusion of growth hormone (30 ng·kg-¹·min-¹) combined with oral placebo
  Interventions: Drug: Growth Hormone, Human; Dietary Supplement: Oral placebo drink
- Saline infusion + oral ketone supplement (Experimental): Participants receive an intravenous saline infusion combined with oral ketone supplementation.
  Interventions: Dietary Supplement: Oral ketone supplement (KetoAid®, KE4); Drug: Saline infusion (placebo)
- Saline infusion + oral placebo (Placebo Comparator): Participants receive a continuous intravenous infusion of saline combined with oral placebo
  Interventions: Drug: Saline infusion (placebo); Dietary Supplement: Oral placebo drink

INTERVENTIONS:
Drug: Growth Hormone, Human — Continuous intravenous infusion of growth hormone (30 ng·kg-¹·min-¹) for approximately 7 hours to induce physiological lipolysis.
  Arms: GH infusion + oral ketone supplement; GH infusion + oral placebo
Dietary Supplement: Oral ketone supplement (KetoAid®, KE4) — Oral administration of D-β-hydroxybutyrate ester (R-1,3-butanediol β-hydroxybutyrate).
  Arms: GH infusion + oral ketone supplement; Saline infusion + oral ketone supplement
Drug: Saline infusion (placebo) — Continuous IV infusion of isotonic saline as placebo for growth hormone.
  Arms: Saline infusion + oral ketone supplement; Saline infusion + oral placebo
Dietary Supplement: Oral placebo drink — Oral administration of an isocaloric placebo drink.
  Arms: GH infusion + oral placebo; Saline infusion + oral placebo

SUMMARY:
KETO-SENSE is a clinical research study investigating how ketone bodies affect energy metabolism and insulin sensitivity in humans. Ketone bodies are naturally produced by the liver during fasting or prolonged exercise and can serve as an alternative fuel for the brain, heart, and muscles.

In this study, ten overweight but otherwise healthy adults aged 55-70 years will participate in four study days at Aarhus University Hospital. Participants will receive one of four interventions in a randomized crossover design: 1) growth hormone (GH) and a ketone supplement, 2) GH and placebo, 3) a saline infusion with the ketone supplement, or 4) placebo (saline infusion and placebo supplement). The study uses advanced PET/CT imaging, indirect calorimetry, and tissue biopsies to measure how ketones influence fat breakdown, glucose uptake, and energy expenditure.

By understanding these mechanisms, the study aims to clarify whether oral ketone supplementation can improve insulin sensitivity and energy metabolism - findings that could be relevant for common conditions such as overweight, insulin resistance, and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 55-70 yr
* BMI: 25 - 35 kg/m2

Exclusion Criteria:

- Any evidence of acute or chronic illnesses, apart from well-controlled hypertension, that is judged by the investigators to impact the study

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Insulin-stimulated glucose uptake in skeletal muscle and organs measured by [¹⁸F]-FDG PET | During four experimental study days conducted over approximately 12 weeks
  Quantification of insulin-stimulated glucose uptake rates in skeletal muscle and selected organs using dynamic [¹⁸F]-FDG PET during a hyperinsulinemic-euglycemic clamp to assess insulin sensitivity.
Tissue-specific uptake of β-hydroxybutyrate and palmitate measured by PET/CT imaging | During four experimental study days conducted over approximately 12 weeks
  Quantification of tissue-specific uptake of β-hydroxybutyrate (BHB) and palmitate in skeletal muscle, adipose tissue, and myocardium using dynamic PET/CT imaging with [¹¹C]-OHB and [¹¹C]-palmitate tracers.
Tissue-specific oxidation of β-hydroxybutyrate and palmitate measured by PET/CT imaging | During four experimental study days conducted over approximately 12 weeks
  Quantification of oxidation rates of β-hydroxybutyrate (BHB) and palmitate in skeletal muscle, adipose tissue, and myocardium using dynamic PET/CT imaging with [¹¹C]-OHB and [¹¹C]-palmitate tracers to assess tissue-specific substrate utilization.
Energy expenditure | During four experimental study days conducted over approximately 12 weeks
  Measurement of resting and insulin-stimulated energy expenditure using indirect calorimetry and analysis of respiratory exchange ratio (RER).
Cardiac output measured by PET/CT imaging | During four experimental study days conducted over approximately 12 weeks
  Quantification of cardiac output in the basal state and during the hyperinsulinemic-euglycemic clamp using dynamic PET/CT imaging to evaluate hemodynamic effects of GH and β-hydroxybutyrate.
Myocardial glucose and fatty acid uptake rates | During four experimental study days conducted over approximately 12 weeks
  Assessment of myocardial substrate metabolism using dynamic PET/CT imaging with [¹⁸F]-FDG and [¹¹C]-palmitate tracers during the basal period and the hyperinsulinemic-euglycemic clamp to quantify myocardial utilization of glucose and fatty acids.

SECONDARY OUTCOMES:
Skeletal muscle pyruvate dehydrogenase (PDHa) enzymatic activity | During four experimental study days conducted over approximately 12 weeks
  Assessment of skeletal-muscle PDHa enzymatic activity determined from the rate of acetyl-CoA production using a radioactivity-based assay and normalized to creatine content in the muscle homogenate.
Adipose tissue lipoprotein lipase (LPL) enzymatic activity | During four experimental study days conducted over approximately 12 weeks
  Determination of heparin-releasable LPL activity in subcutaneous adipose-tissue and muscle biopsies using the glycerol-stabilized method to evaluate triglyceride-derived fatty-acid uptake.
Expression levels of lipolytic regulatory proteins in adipose tissue | During four experimental study days conducted over approximately 12 weeks
  Expression of regulators of lipolysis to assess GH- and BHB-mediated effects on lipid metabolism.
Phosphorylation levels of insulin-regulated proteins in skeletal muscle | During four experimental study days conducted over approximately 12 weeks
  Quantification of phosphorylation levels of insulin-regulated proteins in skeletal-muscle biopsies.
Expression levels of insulin-regulated proteins in skeletal muscle | During four experimental study days conducted over approximately 12 weeks
  Quantification of protein expression levels of insulin-regulated proteins in skeletal-muscle biopsies.
Expression levels of GH-regulated proteins (GHR, JAK2, STAT5, BCL6) in skeletal muscle and adipose tissue | During four experimental study days conducted over approximately 12 weeks
  Quantification of GH-regulated proteins (GHR, JAK2, STAT5, BCL6) in muscle and adipose biopsies using capillary electrophoresis immunoassay for each intervention condition.
Relative mRNA expression of GH-responsive genes (SOCS1-3, CISH, IGF-I) in skeletal muscle and adipose tissue | During four experimental study days conducted over approximately 12 weeks
  Quantification of GH-responsive gene expression (SOCS1-3, CISH, IGF-I) in muscle and adipose biopsies using RT-PCR. Relative mRNA expression will be reported as fold change for each intervention condition.
Skeletal muscle mitochondrial oxidative phosphorylation capacity | During four experimental study days conducted over approximately 12 weeks
  Assessment of mitochondrial oxidative phosphorylation capacity in permeabilized muscle fibers obtained from vastus lateralis biopsies, measured by high-resolution respirometry (Oroboros Oxygraph-2k).
Muscle glycogen content | During four experimental study days conducted over approximately 12 weeks
  Measurement of skeletal-muscle glycogen stores to assess substrate utilization and glucose storage during growth-hormone and ketone interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the small sample size, risk of indirect participant identification, and national data protection regulations (GDPR and Danish Data Protection Act). Aggregated and anonymized summary data will be available upon reasonable request.